CLINICAL TRIAL: NCT02992990
Title: A Prospective Study To Assess Whether A Preoperative Tumor Biopsy Can Improve Upon The Endoscopic Impression Determination Of Stage And Grade In Non-Muscle-Invasive Urothelial Carcinoma Of The Bladder
Brief Title: Bladder Tumor Biopsy Study to Improve Preoperative Determination of Stage and Grade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Guilherme Godoy, Assistant Professor of Urology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-40414
Record Dates: First submitted 2016-12-08; First posted 2016-12-14 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder tumor biopsy (Other): All subjects will undergo a bladder tumor biopsy followed by transurethral resection.
  Interventions: Procedure: Bladder tumor biopsy

INTERVENTIONS:
Procedure: Bladder tumor biopsy — Bladder tumor biopsy performed at the time of the preoperative office flexible cystoscopic evaluation.

SUMMARY:
To assess whether the addition of a bladder tumor biopsy improves the level of agreement between the pretreatment endoscopic impression and the final postoperative pathology determination of stage and grade in non-muscle-invasive urothelial carcinoma of the bladder.

DETAILED DESCRIPTION:
Non-invasive bladder cancer is challenging to treat because it is a condition characterized by frequent recurrences that lead to numerous invasive procedures for detection and treatment. The mainstay of therapy for non-muscle invasive bladder cancer, which has remained unchanged for decades, relies on surgical resection (TUR) associated with utilization of intravesical immunotherapy and chemotherapy. Despite our best efforts, these tumors continue to have suboptimal rates of recurrence and require long-term follow-up with costly and invasive procedures. The rationale for this study is to show that the preoperative biopsy, taken at the time of the office cystoscopic evaluation, improves pre-TUR staging and grading correlation with the final pathology of the resection. Indirectly, this will suggest that the routine use of pre-TUR biopsy provides more accurate information for intraoperative decision-making that can ultimately lead to better management of these patients with non-muscle-invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or females, age 21 or older;
* Clinical evidence of urothelial carcinoma of the bladder;
* Clinically (endoscopic, by physical examination, and/or axial-imaging) deemed non-muscle-invasive tumor of the bladder (cTis-Ta-T1), of any grade, single or multiple, at initial occurrence or recurrent with >12 months interval free of disease;
* Surgically eligible for the TUR;
* Patient or authorized proxy needs to have signed the informed consent form.

Exclusion Criteria:

* History of any muscle-invasive or non-organ confined bladder tumors (T2 or higher);
* Patients with sessile appearing bladder tumors, which may be T2 or higher stage;
* Diagnosis of urothelial carcinoma involving the prostatic urethra or upper urinary tract;
* Concurrent use of anticoagulation medication or chronic use of NSAIDs, including aspirin (other than cardio protective doses of 80mg daily) that has not been appropriately interrupted before the office cystoscopic evaluation;
* Patient deemed medically or psychologically unfit for the surgical procedure;
* Subject has received any investigational medication within 30 days prior to the registration or is scheduled to receive an investigational drug during the course of the study;

Women Exclusion

* Pregnant or lactating women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the kappa agreement score between preoperative and postoperative assessment of stage and grade in non-muscle-invasive bladder tumors. | 3 years
  Assessment of grade, which is the main endpoint will be dichotomous defining lesions between low versus high grade. Stage classification of non-muscle-invasive papillary lesions is also dichotomous between Ta and T1 lesions. CIS can be annotated, but since these are flat, diffuse and non "resectable" in the bladder, they are not part of our main analysis, endpoints, or sample size calculations. The only exception is when the presence of CIS is used to determine grade (high-grade lesion).

CONTACTS AND LOCATIONS:
Overall Officials: Guillherme Godoy, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No